CLINICAL TRIAL: NCT00232791
Title: A Randomized Study With the CYPHER SELECT™ Sirolimus-Eluting Balloon-Expandable Coronary Stent in the Treatment of Patients With de Novo Native Coronary Artery Lesions.
Brief Title: The Study to Compare Cypher Versus Cypher Select in Treating Cornary Artery Lesions.
Acronym: DOMINO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Director Clinical Affairs, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC03-04
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CYPHER SELECT™ Sirolimus-eluting Coronary Stent
  Interventions: Device: Cypher Select
- 2 (Active Comparator): CYPHER™ Sirolimus-eluting Coronary Stent
  Interventions: Device: Cypher

INTERVENTIONS:
Device: Cypher Select — CYPHER SELECT™ Sirolimus-eluting Coronary Stent
  Other Names: PTCA
  Arms: 1
Device: Cypher — CYPHER™ Sirolimus-eluting Coronary Stent
  Other Names: PTCA
  Arms: 2

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the CYPHER SELECT™ Sirolimus-eluting Coronary Stent in reducing angiographic in-stent late loss in de novo native coronary lesions as compared to the CYPHER ™ Sirolimus-eluting Coronary Stent.

DETAILED DESCRIPTION:
This is a multicenter (up to 10 sites), open, prospective, 2-arm, unbalanced, randomized study designed to assess the safety and effectiveness of the CYPHER SELECT™ Sirolimus-eluting Coronary Stent as compared to the CYPHER™ Sirolimus-eluting Coronary Stent. A total of 100 patients will be entered in the study and will be randomized on a 2:1 basis to the CYPHER SELECT™ stent or the CYPHER™ stent. 100 patients with de novo native coronary artery lesions <23 mm in length and more than 2.5 to less than 3.5 mm in diameter by visual estimate who meet all eligibility criteria will be either randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;
2. Single treatment of de novo lesion in a coronary artery which can be appropriately covered by a study stent up to 23mm in length in patients with single or multivessel disease; patients with multiple lesions can be included only if the other lesions are successfully treated before the target lesion;
3. Target lesion is more than 2.5 and less than 3.5mm in diameter (visual estimate);
4. Target lesion is located in a native coronary artery with a maximum lesion length that can be adequately covered by a single 23 mm stent;
5. Target lesion stenosis is > 50% and < 100% (visual estimate).

Exclusion Criteria:

1. A Q-wave or non-Q-wave myocardial infarction within the preceding 72 hours unless the CK and CK-MB enzymes are back to normal;
2. Unprotected left main coronary disease with more than 50% stenosis;
3. Significant (>50%) stenoses proximal or distal to the target lesion that might require revascularization or impede runoff;
4. Have an ostial target lesion;
5. Angiographic evidence of thrombus within target lesion;
6. Calcified lesions which cannot be successfully predilated;
7. Ejection fraction less than 30%;
8. Totally occluded vessel (TIMI 0 level);
9. Direct Stenting;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2004-01; Primary Completion 2004-08 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Angiographic in-stent late loss | 6 months

SECONDARY OUTCOMES:
In-stent mean percent diameter stenosis | anytime post-procedure
In-target vessel segment MLD | 6 months
In-stent MLD | 6 months
Target Lesion Revascularization (TLR) | 6 months
Target Vessel Revascularization (TVR) | 6 months
Major Adverse Cardiac Events (MACE) | 30 days, 6 and 12 months
In-stent volume of restenosis determined by IVUS | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: R. H. Stables, MD, Principal Investigator — Cardiothoracic Centre Liverpool
Locations (1):
- Cardiothoracic Center Liverpool, Liverpool, United Kingdom